CLINICAL TRIAL: NCT02732054
Title: Comparison of Immunogenicity and Safety of 4 Standard Doses and 3 Standard Doses of Hepatitis B Vaccination in HIV-infected Adults Who Have CD4 < 200 Cells/mm3
Brief Title: Hepatitis B Vaccination in HIV-infected Adults With Low CD4 Cell Counts
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Romanee Chaiwarith, Associate Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Research ID: 02891
Record Dates: First submitted 2016-03-31; First posted 2016-04-08 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Hepatitis B
Keywords: HBV vaccination, immunity
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIV-Group 1 (Active Comparator): Receiving three intramuscular injections of 20 µg of recombinant hepatitis B vaccine [(CIGB) La Habana, Cuba] at months 0, 1, and 6
  Interventions: Biological: Recombinant Hepatitis B vaccine [(CIGB) La Habana, Cuba]
- HIV-Group 2 (Experimental): Receiving four intramuscular injections of 20 µg of recombinant hepatitis B vaccine [(CIGB) La Habana, Cuba] at months 0, 1, 2, and 6
  Interventions: Biological: Recombinant Hepatitis B vaccine [(CIGB) La Habana, Cuba]

INTERVENTIONS:
Biological: Recombinant Hepatitis B vaccine [(CIGB) La Habana, Cuba] — Different HBV vaccine regimen in each group

SUMMARY:
This study aimed to evaluate the efficacy of different hepatitis B vaccination regimens in HIV-infected adults with low CD4 cell count in northern Thailand.

DETAILED DESCRIPTION:
HIV-infected adults with CD4+ cell counts < 200 cells/mm3, undetectable plasma HIV-1 RNA, and negative for all HBV markers were randomly assigned to receive one of these 2 regimens of recombinant hepatitis B vaccine (Centro De Ingenieria Genetica Y Biotecnologia, La Habana, Cuba); 1) 20 μg IM at months 0, 1, and 6 (3-standard doses group), and 2) 20 μg IM at months 0, 1, 2, 6 (4-standard doses group).

This study aimed to evaluate the efficacy and safety of these 2 hepatitis B vaccination regimens at month 7 after vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infection
2. ≥18 years old
3. Received combination antiretroviral therapy for at least 1 year
4. Had a CD4+ cell count < 200 cells/mm3 for at least 1 year
5. Undetectable plasma HIV-1 RNA for at least 1 year
6. Negative for hepatitis B surface antigen (HBsAg), antibody to hepatitis B surface antigen (anti-HBs), and antibody to hepatitis B core antigen (anti-HBc),
7. Had no history of previous HBV vaccine
8. Negative for antibody to hepatitis C virus (anti-HCV)
9. No active opportunistic infections (at the time of screening)
10. Willing to sign an informed consent
11. Able to return for follow-up.

Exclusion criteria

1. Pregnancy or lactation
2. History of hypersensitivity to any component of the vaccine
3. Active malignancy receiving chemotherapy or radiation, or other immunocompromised conditions besides HIV (e.g., solid organ transplant), received immunosuppressive (e.g., corticosteroid ≥ 0.5 mg/kg/day) or immunomodulating treatment in the last six months before screening visit
4. Renal insufficiency (creatinine clearance <30 mL/min)
5. Decompensated cirrhosis (Child-Pugh class C)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with protective immunity against HBV | 1 month after vaccination
  comparison of proportion of participants who had protective immunity (anti-HBS titer >=10 mIU/ml) against HBV between HIV group 2 v.s. HIV group 1

SECONDARY OUTCOMES:
The geometric means of anti-HBs titers | 1 month after vaccination
  Comparison of the geometric means of anti-HBS titers between HIV group 2 v.s. HIV group 1
Proportion of participants with high level of immune response against HBV | 1 month after vaccination
  Comparison of proportion of participants who had anti-HBS titers >= 100 mIU/ml between HIV group 2 v.s. HIV group 1

CONTACTS AND LOCATIONS:
Overall Officials: Romanee Chaiwarith, MD, Principal Investigator — Thailand Maharaj Nakorn Chiang Mai Hospital, Department of Medicine, Chiang Mai University Muang, Chiang Mai Thailand
Locations (1):
- Maharaj Nakorn Chiang Mai Hospital, Department of Medicine, Chiang Mai University, Muang, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No